CLINICAL TRIAL: NCT07348042
Title: An Open, Multi-center Phase I Clinical Study Evaluating the Safety, Tolerance, Pharmacokinetics and Immunogenicity of RGL-270 Single Drug and Combined With Adebelimab in Patients at High Risk of Recurrence After Radical Treatment of Malignant Solid Tumors
Brief Title: Study of RGL-270 Single Drug and Combined With Adebelimab in Patients in Patients at High Risk of Recurrence After Radical Treatment of Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xian-Jun Yu (Other)
Responsible Party: Sponsor-Investigator, Xian-Jun Yu, The current director of Fudan University Affiliated Cancer Hospital and the director of Shanghai and Fudan University Pancreatic Tumor Research Institute., Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGL-270-101
Record Dates: First submitted 2025-05-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Tumor, Solid
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Increase the dose of single-drug treatment (Experimental): (Part A)
  Interventions: Drug: RGL-270 Injection
- Combined treatment dose increase (Experimental): (Part B)
  Interventions: Drug: RGL-270 Injection; Drug: Adebelimab Injection
- Combined treatment dose expansion (Experimental): (Part C)
  Interventions: Drug: RGL-270 Injection; Drug: Adebelimab Injection

INTERVENTIONS:
Drug: RGL-270 Injection — Repeated medication, increase the dose
Drug: Adebelimab Injection — Repeated medication, the dose is maintained
  Arms: Combined treatment dose expansion; Combined treatment dose increase

SUMMARY:
This study is a phase I clinical trial of multi-center, open label, dose increase and dose expansion. It aims to evaluate the safety, tolerance, PK characteristics, immunogenicity and initial efficacy of personalized new antigen mRNA vaccine RGL-270 (hereinafter referred to as RGL-270) alone and combined with adebelizumab in patients with high risk of recurrence of malignant solid tumors after radical treatment.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening period

1. Subjects should understand and abide by the relevant research procedures, and voluntarily sign the prior informed consent form;
2. Age 18-75 years old (including boundary value), gender is not limited;
3. For malignant solid tumors confirmed by histology or cytology after radical resection, the subjects are allowed to complete standard adjuvant treatment, or no standard adjuvant treatment, or adjuvant treatment intolerance before receiving the first administration of this study:
4. Willing to provide sufficient tumor tissue specimens and peripheral blood for genetic testing and new antigen analysis;
5. Fertile female subjects and male subjects whose partners are women of childbearing age must agree to comply with the contraceptive requirements for 6 months from the signing of the pre-informed consent form until the end of the last treatment.

Screening period

1. Subjects should understand and abide by the relevant research procedures, and voluntarily sign the owner's informed consent form;
2. Eastern American Oncology Collaborative Group (ECOG) score: 0 or 1 point;
3. Willing to provide blood samples needed to detect immunogenicity and biomarkers before and after drug treatment;
4. The functions of important organs meet the following criteria (no blood components and cell growth factors have been used within 14 days before the start of research and treatment):

   A) Blood routine: neutrophil count (ANC) ≥1.5×109/L, lymphocyte count (LYM) ≥0.5×109/L, platelet count (PLT) ≥1× normal lower limit (LLN), hemoglobin (Hb) ≥90g/L; B) Blood biochemical: total bilirubin (TBIL) ≤1.5× normal upper limit (ULN), glutathione transaminase (ALT) and glutathione transaminase (AST) ≤2.5×ULN, serum albumin (ALB) ≥30g/L, serum creatine (Scr) ≤1×ULN; C) Coagulation routine: International Standardized Ratio (INR) ≤1.5, activated partial prothrombin time (APTT) ≤1.5×ULN; D) Heart function: Left ventricular blood ejection fraction (LVEF) ≥50%; E) Electrocardiogram: The QT interval (QTcF) corrected by Fridericia method is <470 milliseconds; the QTc interval must be corrected according to Fridericia's standard, and the correction formula QTcF=QT/RR^0.33.
5. Clinical examination, chest and abdomen CT and head MRI baseline radiological evaluation within 14 days before the first vaccine administration showed no evidence of disease recurrence;
6. Fertile female subjects must take a serum pregnancy test within 7 days before the first vaccination, and the result is negative and must be non-lactating.

Exclusion Criteria:

* Pre-screening period

  1. Have received immune cell or tumor vaccine treatment, including but not limited to tumor infiltration lymphocytes (TILs), chimeric antigen receptor T cells (CAR-T), T cell receptor chimeric T cells (TCR-T) and therapeutic tumor vaccines;
  2. Plan to inoculate live attenuated vaccine during the screening period or during the research period and within 90 days after the end of the research drug treatment (inactivated vaccine is allowed);
  3. Anyone who is evaluated by researchers as not suitable for immunotherapy;
  4. There is an autoimmune disease (except for hypothyroidism who need hormone replacement treatment caused by autoimmune thyroiditis);
  5. Known history of epilepsy or other symptomatic neurological diseases;
  6. Known history of psychotropic substance abuse, alcoholism or drug abuse;
  7. There is evidence of active tuberculosis infection within 1 year before the pre-screening period and during the pre-screening period, whether it is treated or not;
  8. Subjects with known or suspected interstitial pneumonia, or evidence of interstitial pneumonia in the chest CT during the pre-screening period; known history of idiopathic pulmonary fibrosis, mechanized pneumonia (such as occlusive bronchitis or occult mechanized pneumonia);
  9. Combined history of other malignant tumors within 5 years before the pre-screening period;
  10. Known history of allogeneic organ transplantation or history of allogeneic hematopoietic stem cell transplantation;
  11. Known allergy to research drugs or any of their auxiliaries, or a history of severe allergic reactions to other vaccines;
  12. Suffering from congenital or acquired immunodeficiencies, such as cellular immunodeficiencies (such as DiGeorge syndrome, T-negative severe combined immunodeficiency [SSCID]) or combined T-cell and B-cell immunodeficiency (such as T- and B-negative combined immunodeficiency, Wiskott-Al Drich syndrome, ataxia telangiectasia, common variable immunodeficiency); or infected with human immunodeficiency virus (HIV);
  13. Poorly controlled or severe cardiovascular and cerebrovascular diseases: congestive heart failure (NYHA standard III or level IV), severe arrhythmia requiring treatment or intervention, and poorly controlled hypertension after full treatment (systolic pressure ≥160mmHg, diastolic pressure ≥100mmHg );
  14. Pregnant or lactating female subjects;
  15. The data analysis results of tumor tissue sequencing show that there are not enough new antigens available for vaccine preparation or vaccine preparation fails;
  16. The researcher judges that the subject may not be able to continue to participate in the study:
* Any other disease in which the subject faces the risk of safety;
* Subjects with poor compliance or active request to withdraw from pre-screening;
* There is a recurrence of the disease during the pre-screening period. Screening period

  1. Postoperative complications have not recovered, or the complications are higher than the Clavien-Dindo complication grade 2;
  2. The toxicity caused by auxiliary treatment before the first vaccine administration has not recovered to the baseline level or >1 (except for hair loss and pigmentation), and the neurotoxicity is >2;
  3. There is evidence of active tuberculosis infection during the screening period, whether it is treated or not;
  4. Chest CT during the screening period suggests evidence of interstitial pneumonia;
  5. Concurrent severe infection within 28 days before the first vaccination (such as intravenous drip of antibiotics, antifungal or antiviral drugs according to clinical diagnosis and treatment standards);
  6. Within 28 days before the first vaccination, there is pleural fluid or ascites that are not clinically controlled and require thoracic puncture or abdominal puncture drainage;
  7. Active hepatitis B (defined as active hepatitis B virus surface antigen [HBsAg] test results during the screening period are positive and HBV DNA≥500IU/mL or higher than the upper limit of the normal detection value of the research center), or hepatitis C (defined as hepatitis C antibodies during the screening period [HCV -Ab] The test result is positive, and HCV-RNA is positive);
  8. Myocardial infarction or stroke occurred within 3 months before the first vaccination (except for transient cerebral ischemia and cavity cerebral infarction), or unstable angina pectoris within 1 month;
  9. Arteriovenous thrombosis, such as deep vein thrombosis or pulmonary embolism, occurred within 3 months before the first vaccination;
  10. The researcher judges other circumstances that may affect the progress of clinical research and the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-09-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of RGL-270 monotherapy or the maximum dose (MAD) when MTD is not reached, and determine the recommended extended dose (RDE) for RGL-270 | Day 1 to week 24 after RGL-270 administration
  Evaluate the safety and tolerability of RGL-270 monotherapy and combined with , Adebelimab in patients at high risk of recurrence after radical treatment of malignant solid tumors, determine the maximum tolerated dose (MTD) of RGL-270 monotherapy or the maximum dose (MAD) when MTD is not reached, and determine the recommended extended dose (RDE) for RGL-270 combined with Adebelimab treatment

SECONDARY OUTCOMES:
Specific T-cell response and antidrug antibody (ADA) | Day 1 to week 24 after RGL-270 administration
  Evaluate the rate of specific T-cell response positivity and change in response from baseline, and the rate and duration of antibody to drug (ADA) positivity
Preliminary therapeutic effect- DFS rate | Day 1 to month 24 after RGL-270 administration
  Evaluate the disease-free survival (DFS), 18-month/24-month DFS rate
Preliminary therapeutic effect- OS rate | Day 1 to month 24 after RGL-270 administration
  Evaluate the overall survival (OS), 18-month/24-month OS rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No